CLINICAL TRIAL: NCT00977028
Title: Tumescent Lidocaine Bioavailability and Absorption Kinetics:Maximum Safe mg/kg Lidocaine Dosage
Brief Title: Tumescent Lidocaine Maximum Safe mg/kg Dosage
Acronym: TLA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Klein, Jeffrey A., M.D. (Individual)
Responsible Party: Jeffrey A. Klein, MD, Jeffrey A. Klein, MD, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1 TLA Peak
Record Dates: First submitted 2009-09-12; First posted 2009-09-15 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Anesthesia
Keywords: Tumescent; Local Anesthesia; Lidocaine; Dosage Maximum; Subcutaneous infiltration; maximum Safe mg per kg dosage of lidocaine; Tumescent Local Anesthesia
MeSH Terms: interventions — Lidocaine; Epinephrine; Anesthesia; Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tumescent Lidocaine with liposuction (Experimental): Determine maximum safe mg/kg dosage of tumescent lidocaine with liposuction
  Interventions: Drug: Tumescent Local Anesthesia (lidocaine, epinephrine); Procedure: Liposuction
- Tumescent Lidocaine No Liposuction (Experimental): Determine maximum safe mg/kg dosage of tumescent lidocaine without liposuction
  Interventions: Drug: Tumescent Local Anesthesia (lidocaine, epinephrine); Procedure: Liposuction

INTERVENTIONS:
Drug: Tumescent Local Anesthesia (lidocaine, epinephrine) — Tumescent solution of lidocaine (up to 1 gm per liter) and epinephrine (up to 1 mg per liter)with subcutaneous infiltration of up to 45 mg per kilogram
  Other Names: Tumescent; Lidocaine; Xylocaine; Epinephrine; Local; Anesthesia
Procedure: Liposuction — Subcutaneous infiltration of tumescent local anesthesia (large volumes of dilute lidocaine and epinephrine) on at least two different occasions, followed by sequential serum samples every two hours for HPLC determination of serum lidocaine concentration and peak serum lidocaine concentration, initially without subsequent liposuction and finally on the last occasion with liposuction
  Other Names: tumescent local anesthesia; lidocaine; epinephrine

SUMMARY:
This pharmacokinetic clinical trial is a dose ranging study of lidocaine in tumescent local anesthesia. The goal is to understand the absorption pharmacokinetic of tumescent lidocaine and to determine an objective (statistical) estimate of the maximum safe mg/kg dosage of lidocaine in tumescent local anesthesia without liposuction.

DETAILED DESCRIPTION:
Background:

Tumescent local anesthesia (TLA) permits a wide variety of therapeutic surgical procedures of subcutaneous tissues and skin to be performed totally by local anesthesia ( ). Infiltration of a sufficient volume of TLA causes the target tissues become temporarily tumescent, or swollen and firm.

TLA is defined as the subcutaneous infiltration of a large volume of a tumescent local anesthetic solution (TLAS). The safe use of TLA requires the safe formulation and safe use of a tumescent local anesthetic solution (TLAS). By definition TLAS contains very dilute lidocaine (≤ 1 gm/liter = 0.1%) and epinephrine (≤ 1 mg/liter = 1:1,000,000) with sodium bicarbonate (10 milliequivalents/liter) in a physiologic crystalloid solution. Bicarbonate, an essential ingredient, neutralizes the acid pH of commercial lidocaine and epinephrine thereby eliminating the intense stinging discomfort which often associated with the infiltration of commercial local anesthetics. Lidocaine which has been infiltrated for TLA is referred to as tumescent lidocaine.

The FDA-approved maximum recommended dosage is 7 mg/kg for lidocaine with epinephrine infiltration local anesthesia. However with TLA much larger mg/kg dosages of lidocaine are used. The safety and efficacy of TLA is based on the unexpected slow lidocaine absorption associated with large volumes of very dilute lidocaine and epinephrine when infiltrated into subcutaneous tissue. Published estimates of a maximum safe mg/kg dosage of tumescent lidocaine are derived from liposuction patients and have ranged from 35 mg/kg to 55 mg/kg ( ) and much higher lidocaine doses without evident toxicity have been reported.

Liposuction, a cosmetic surgical procedure which removes subcutaneous fat, also removes some tumescent lidocaine thereby reducing lidocaine bioavailability. In contrast, therapeutic surgeries usually do not remove subcutaneous lidocaine and therefore the bioavailability of lidocaine is relatively increased as is the peak serum lidocaine concentration (Cmax) and the risk of lidocaine toxicity. Because TLA is now used for surgical procedures unrelated to liposuction, it is desirable to have a reliable estimate of the maximum safe dosage of tumescent lidocaine based on clinical data from subjects not having liposuction.

The goal of the present study is to obtain reliable estimates of the maximum safe mg/kg dosage of lidocaine after tumescent local anesthesia both with and without subsequent liposuction. The plan for the present pharmacokinetic study involves the following steps:

1. Show that there is a significant difference between the bioavailability of tumescent lidocaine with or without liposuction. This will validate the need to determine the maximum safe mg/kg dosage of tumescent lidocaine without liposuction.
2. Show that the magnitude of the peak serum lidocaine concentration is a linear function of the mg/kg dosage of tumescent lidocaine, with and without liposuction. This will support the use of interpolation and extrapolation in the discussion of results.
3. For any specified mg/kg dosage of tumescent lidocaine, estimate the risk that the peak serum lidocaine concentration will exceed the 6 µg/ml toxic threshold.

Methods:

The protocol and consent forms for this research has been approved by an institutional review board. All clinical procedures are to be conducted within an accredited ambulatory surgery center.

Serum lidocaine concentration will be measured by high pressure flame chromatography (HPFC). Female volunteer subjects will each participate in three procedures. Each procedure involves the infiltrating of TLA followed by sequential serum samples obtained from a peripheral vein via plastic catheter at time (T) = 0, 2, 4, 6, 8, 10, 12, 14, 16, 18 and 24 hours to be assayed for lidocaine concentration by HPFC. For each procedure, the mg/kg dosage of tumescent lidocaine and a corresponding peak or maximum serum lidocaine concentration (Cmax) are to be recorded.

The areas targeted for infiltration of tumescent local anesthesia (TLA) will vary from subject to subject and include abdomen, hips, outer thigh, inner thighs and knees, female breasts, lateral thorax and back. For each subject, the first two investigative procedures involve an infiltration of TLA without subsequent liposuction; in the third procedure the subject receive TLA followed by liposuction. Thus each patient serves as her own control. Liposuction will be initiated one to two hour after completion of the infiltration process. For each subject the TLA infiltration will be in the same area and sequential infiltrations are to be separated by at least two weeks. As compensation for participation in the three clinical studies, each procedure requiring more than 24 hours, the patients will receive liposuction of the targeted area at no cost.

The total mg/kg dosage of tumescent lidocaine will vary between patients and for different procedures within the same patient. An individual patient will receive the same mg/kg dosage of tumescent lidocaine on at least two occasions, once followed by liposuction and at least once without liposuction. Some patients will receive the same dosage of tumescent lidocaine for all three procedures. Similarly, in order to explore the effect of varying the concentrations lidocaine or the concentration of epinephrine within the TLA solution or to understand the effect of varying the mg/kg dosage of TLA, in some patients these factors will be varied.

In order to determine if liposuction significantly affects the amount of lidocaine that enters the systemic circulation, the bioavailability associated of tumescent lidocaine without and with liposuction will be compared. The statistical significance of the difference between the area under the curve (AUC) without liposuction and the AUC with liposuction will be calculated For each procedure, a graph of the sequential serum lidocaine concentrations C(T) as a function of time (T) will be drawn and each peak serum lidocaine concentration and time will be recorded both with liposuction and without liposuction. Confidence intervals will be determined in order to estimate the risk that, for any given mg/kg dosage, the Cmax will exceed the toxic threshold for lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female (ASA class 1 or 2)
* Desires liposuction
* Easily accessible veins

Exclusion Criteria:

* History of Hepatitis C, HIV
* ASA class greater or equal to 3

Ages: 18 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-01; Primary Completion 2011-07 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Peak or maximum serum lidocaine concentration (Cmax) following a given mg/kg dosage of lidocaine delivered by subcutaneous infiltration of tumescent local anesthesia | 24 hours

SECONDARY OUTCOMES:
Cmax following 45mg/kg tumescent lidocaine has a Normal distribution. We define the probability that Cmax exceeds 6 microgram/ml, the toxic threshold for lidocaine as a function of lidocaine dosage. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Klein, MD, Principal Investigator — University of Californiia, Riverside
Locations (1):
- Capistrano Surgery Center, San Juan Capistrano, California, United States